CLINICAL TRIAL: NCT02409433
Title: Prospective, Randomized, Single-blinded Comparative Trial of IV Lacosamide Versus Phenytoin for Seizure Management
Brief Title: Comparative Trial of IV Lacosamide Versus Phenytoin for Seizure Management
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: due to slow recruitment and budgetary restraints study was prematurely terminated
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: UCB Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Jorge Burneo, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100739
Record Dates: First submitted 2015-04-01; First posted 2015-04-06 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Seizures
Keywords: lacosamide; phenytoin
MeSH Terms: conditions — Seizures | interventions — Lacosamide; Phenytoin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- lacosamide (Experimental): The lacosamide group will receive a loading dose of 400 mg IV, and on maintenance dose of up to 400 mg every 12 hours.
  Interventions: Drug: lacosamide
- phenytoin (Active Comparator): the phenytoin group will receive a loading dose of 20 mg/K IV, maximum of 2000 mg, given over 60 min. and will be started on a maintenance dose of 5 mg/K/day. Levels will be checked accordingly.
  Interventions: Drug: Phenytoin

INTERVENTIONS:
Drug: lacosamide — Comparison of patients treated with IV lacosamide to those treated with phenytoin in the intensive care unit setting.
  The lacosamide group will receive a loading dose of 400 mg IV, and on maintenance dose of up to 400 mg every 12 hours.
  Other Names: Vimpat
  Arms: lacosamide
Drug: Phenytoin — the phenytoin group will receive a loading dose of 20 mg/K IV, maximum of 2000 mg, given over 60 min. and will be started on a maintenance dose of 5 mg/K/day.
  Other Names: Dilantin
  Arms: phenytoin

SUMMARY:
The Investigator plans to perform a prospective, randomized, single blinded, study that will compare patients treated with IV lacosamide to those treated with Phenytoin in the Intensive Care Unit (ICU) setting. The investigator will also evaluate the rate of clinically evident and sub-clinical seizures, and to compare long-term outcomes between patients treated with lacosamide and those treated with Phenytoin.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic Brain Injury (TBI) or Subarachnoid hemorrhage (SAH)
* Admitted to the hospital less than 48 hours prior to randomization
* Glasgow Coma Scale (GCS) score 3-8 (inclusive), or GCS motor score of five or less and abnormal CT scan showing intracranial pathology
* Hemodynamically stable
* Older than 18 years of age

Exclusion Criteria:

* No IV access
* Spinal cord injury
* History of or CT confirmation of previous brain injury, including brain tumor, stroke, or a spontaneous intracerebral hemorrhage
* Hemodynamically unstable
* Suspected anoxia
* Liver failure
* Younger than 18 years of age
* Pregnant
* Allergy to phenytoin or lacosamide
* Inability to obtain consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Clinical Adverse Events | 6 months
  Safety: the primary outcome measure will be the incidence of clinical adverse events. Patients will be evaluated daily during the hospital stay for seizures, fever, neurological changes, cardiovascular, hematologic and dermatologic abnormalities, liver failure, renal failure, and death. Each adverse event will be classified by the principal investigator as attributable or possibly attributable to the study drug versus other events. Serious adverse events for these to study will be defined as those that result in death, prolonged hospitalization, life threatening events, persistent or significant disability, or an important medical event that may not be immediately life threatening or result in death but based upon appropriate medical judgment may jeopardize the participant, or may require medical or surgical intervention to prevent one of the other outcomes listed.

SECONDARY OUTCOMES:
Efficacy | 6 months
  Efficacy: the secondary endpoints will be seizure frequency and long-term outcomes (measure by disability scales). All patients will be monitored on continuous EEG for 72 hours or until a week and following commands. Since over 50% of initial seizure activity in these patients are usually subclinical as reported in the finished studies, and about 90% of the seizures happen within the first two days of admission to the ICU, the investigator would stop EEG recordings once patient awake, or by 72 hours after admission if there were no seizures.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Burneo, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- University Hospital, London, Ontario, Canada